CLINICAL TRIAL: NCT01567644
Title: Clinical Trial Evaluating the Treatment of Patients With Refractory Chronic Angina Pectoris With Low Intensity Extracorporeal Shockwave Therapy Device
Brief Title: Extracorporeal Shockwave Therapy for the Treatment of Refractory Chronic Angina Pectoris
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medispec (Industry)
Collaborators: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESMR-NRW-DE
Record Dates: First submitted 2010-11-15; First posted 2012-03-30 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Refractory Angina Pectoris
Keywords: Extracorporeal Shockwave Therapy; Myocardial Ischemia; Refractory Angina
MeSH Terms: conditions — Angina Pectoris; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Shockwave Therapy (Experimental): Patients in this group receive shockwave therapy.
  Interventions: Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec)

INTERVENTIONS:
Device: Cardiac Extracorporeal Shockwave Therapy generator (Cardiospec) — Energy Density - 0.09 mJ/mm2
  Other Names: Cardiospec; ESMR therapy; Extracorporeal Shockwave Myocardial Revascularization

SUMMARY:
Low intensity shockwaves have been proven in animal studies to induce local growth of new blood vessels from existing ones.

The hypothesis of this study is that shockwave therapy could improve the symptoms of patients with refractory angina not amenable to revascularization with angioplasty or bypass surgery.

DETAILED DESCRIPTION:
Low intensity shockwaves (1/10 the ones used in Lithotripsy) are delivered to myocardial ischemic tissue. Shockwaves are created by a special generator and are focused using a shockwave applicator device. The treatment is guided by standard echocardiography equipment. The shockwaves are delivered in synchronization with Patient R-wave to avoid arrhythmias. The treatment is painless.

At first, the patient undergoes stress- PET testing to identify the ischemic areas. Following that, the same area is localized by the ultra-sound device and the shockwaves are focused to the ischemic area. Several treatments are required for optimal results.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic stable angina pectoris.
* Documented myocardial segments with reversible ischemia
* AP CCS class of III-IV.
* Stable dosage of medication used to treat angina for at least 6 weeks prior to enrollment.
* Exercise tolerance time < 10 min (modified Bruce)
* Two ETT tests results (within two weeks) averaging no more than 25% of their mean
* Documented epicardial coronary artery disease not amenable to angioplasty or CABG.
* Signed an IRB approved informed consent form.
* Life expectancy of > 12 months.

Exclusion Criteria:

* Intraventricular thrombus
* Malignancy in the area of treatment
* Severe COPD
* No smoking during the study procedure
* MI less < 3 months prior to treatment
* Severe Valvular disease
* Child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2008-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Change in AP-CCS | 6 Months
  The AP CCS Stage at the 6 months post baseline.

SECONDARY OUTCOMES:
Exercise tolerance time | 6 Months
  The change in Total Exercise Time (Exercise Tolerance Test-ETT) from baseline to 6 months post baseline
Change in PET scan | 6 months
  The change in perfusion in pharmacological induced stress PET scan (at rest and at stress) from baseline to 6 months post baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Faber, Prof. MD, Principal Investigator — Heart and Diabetes Center North-Rhine Westfalia
Locations (1):
- Heart and Diabetes Center North-Rhine Westfalia, Bad Oeynhausen, Germany